CLINICAL TRIAL: NCT01414855
Title: A Phase II, Open-Label, Multicenter Study of Efficacy, Safety, and Biomarkers in Patients With Previously Untreated Advanced Diffuse Large B-Cell Lymphoma Treated With GA101 (RO5072759) in Combination With CHOP Chemotherapy
Brief Title: A Study of Obinutuzumab [RO5072759 (GA101)] in Combination With CHOP Chemotherapy in Patients With Previously Untreated Advanced Diffuse Large B-Cell Lymphoma (GATHER)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAO4915g
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — obinutuzumab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- obinutuzumab + CHOP (Experimental): Participants received 1000 mg obinutuzumab intravenously on Day 1 of each 21-day cycle for 8 cycles; during Cycle 1 administration also on Days 8 and 15. Participants also received standard CHOP therapy (cyclophosphamide, doxorubicin, vincristine and prednisone) for 6 cycles.
  Interventions: Drug: obinutuzumab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone; Drug: vincristine

INTERVENTIONS:
Drug: obinutuzumab — 1000 mg intravenously on Day 1 of each 21-day cycle, 8 cycles; during Cycle 1 administration also on Days 8 and 15.
Drug: cyclophosphamide — 750 mg/m^2 intravenous (IV), Day 1 of each 21-day cycle, 6 cycles.
Drug: doxorubicin — 50 mg/m^2 IV, Day 1 of each 21-cycle, 6 cycles.
Drug: prednisone — 100 mg/day, Days 1 through 5 of each 21-day cycle, 6 cycles.
Drug: vincristine — 1.4 mg/m^2 IV, Day 1 of each 21-day cycle, 6 cycles.

SUMMARY:
This open-label, multicenter study will evaluate the efficacy and safety of obinutuzumab [RO5072759 (GA101)] in combination with CHOP (Cyclophosphamide, Doxorubicin, Vincristine, Prednisone) chemotherapy in patients with advanced diffuse large B-cell lymphoma. Patients will receive 8 cycles of obinutuzumab (1000 mg intravenously on Day 1 of each 21-day cycle, during Cycle 1 obinutuzumab will also be infused on Days 8 and 15) in combination with CHOP chemotherapy on Day 1 of cycles 1 to 6. A substudy will investigate the drug-drug interaction of obinutuzumab with CHOP chemotherapy agents. For the substudy, an additional cohort of approximately 15 patients are planned to be enrolled at a subset of investigational sites.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years of age
* Previously untreated cluster of differentiation antigen 20 (CD20)-positive diffuse large B-cell lymphoma
* Ann Arbour Stage III/IV and bulky II (mass >10 cm)
* At least one bi-dimensionally measurable lesion defined as >1.5 cm in its largest dimension by CT scan
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Left ventricular ejection fraction ≥50%
* Adequate hematologic function

Exclusion Criteria:

* Transformed lymphoma (follicular IIIB) if previously treated with chemotherapy or immunotherapy
* Prior therapy for diffuse large B-cell lymphoma except for nodal biopsy or local irradiation
* Central nervous system (CNS) lymphoma, primary mediastinal large cell lymphoma, primary cutaneous lymphoma, primary effusion lymphoma
* Patients who received cytotoxic drugs or rituximab as part of their treatment for another condition (e.g. rheumatoid arthritis) or prior use of an anti-CD20 antibody
* Chemotherapy or other investigational therapy within 28 days prior to the start of Cycle 1
* Contraindication to any of the individual components of CHOP, including prior receipt of anthracyclines
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* History of other malignancy, except for curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix, or malignancy treated with or without curative intent and in remission without treatment for ≥2 years prior to enrolment
* Positive for hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or human T-cell leukemia virus (HTLV-1) infection
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08-31 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2016-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (38):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - cCare, Encinitas, California
  - University of Colorado Cancer Center Department of Hematology, Aurora, Colorado
  - Rocky Mountain Cancer Ctr - Denver (Williams), Denver, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Florida Cancer Specialists; Department of Oncology, Fort Myers, Florida
  - Florida Cancer Specialists; Saint Petersburg, St. Petersburg, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Northwestern University; Robert H. Lurie Comp Can Ctr, Chicago, Illinois
  - Onc Hem Assoc of Central IL, Peoria, Illinois
  - McFarland Clinic, Ames, Iowa
  - Jewish Cancer Care, Louisville, Kentucky
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - MT Cancer Inst Fndtn; MT Can Spec, Missoula, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - MSKCC at Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Memorial Sloan-Kettering; Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSKCC at Mercy Med Ctr, Rockville Centre, New York
  - MSKCC at Sleepy Hollow, Sleepy Hollow, New York
  - Emerywood Hematology and Onc, High Point, North Carolina
  - Willamette Valley Cancer Insitute and Research Center, Springfield, Oregon
  - Medical University of SC (MUSC), Charleston, South Carolina
  - SCRI-Tennessee Oncology, Nashville, Tennessee
  - Onc & Hem Assoc; USO Cent Pharm, Fort Worth, Texas
  - MD Anderson Cancer Center Department of Lymphoma & Myeloma, Houston, Texas
  - Methodist Hospital Research Institute, Houston, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas
  - USO - Tyler Cancer Ctr, Tyler, Texas
  - Blue Ridge Cancer Care - Roanoke, Roanoke, Virginia
  - Medical Oncology Associates, Spokane, Washington
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Aurora Bay Care Medical Center, Green Bay, Wisconsin

REFERENCES:
- [Derived] Gibiansky E, Gibiansky L, Buchheit V, Frey N, Brewster M, Fingerle-Rowson G, Jamois C. Pharmacokinetics, exposure, efficacy and safety of obinutuzumab in rituximab-refractory follicular lymphoma patients in the GADOLIN phase III study. Br J Clin Pharmacol. 2019 Sep;85(9):1935-1945. doi: 10.1111/bcp.13974. Epub 2019 Jul 12. PMID 31050355
- [Derived] Sharman JP, Forero-Torres A, Costa LJ, Flinn IW, Inhorn L, Kelly K, Bessudo A, Fayad LE, Kaminski MS, Evens AM, Flowers CR, Sahin D, Mundt KE, Sandmann T, Fingerle-Rowson G, Vignal C, Mobasher M, Zelenetz AD. Obinutuzumab plus CHOP is effective and has a tolerable safety profile in previously untreated, advanced diffuse large B-cell lymphoma: the phase II GATHER study. Leuk Lymphoma. 2019 Apr;60(4):894-903. doi: 10.1080/10428194.2018.1515940. Epub 2018 Oct 2. PMID 30277102

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obinutuzumab + CHOP
Started | 100
Completed | 71
Not Completed | 29
Not completed — Death | 17
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Groups:
- Obinutuzumab + CHOP: Participants received 1000 mg obinutuzumab intravenously on Day 1 of each 21-day cycle for 8 cycles; during Cycle 1 administration also on Days 8 and 15. Participants also received standard CHOP therapy for 6 cycles.
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate as Assessed by the Investigator at the End of Treatment
Description: Complete response rate is defined as the percentage of participants with Complete Response (CR) according to the Revised Response Criteria for Malignant Lymphoma (Cheson et al., 2007). Disease response was evaluated by the investigator using regular clinical and laboratory examinations, fluorodeoxyglucose-positron emission tomography (FDG-PET) and computed tomography (CT). CR is the disappearance of all evidence of disease.
Time Frame: From the first dose of study treatment to end of treatment response assessment (approximately 228 to 258 days)
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
percentage of participants | 55.0 [44.73 to 64.97]

2. Primary Outcome: Overall Response Rate (ORR) as Assessed by the Investigator at the End of Treatment
Description: Overall response rate was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) according to the Revised Response Criteria for Malignant Lymphoma (Cheson et al., 2007). Disease response was evaluated by the investigator using regular clinical and laboratory examinations, FDG-PET and computed tomography (CT). CR is the disappearance of all evidence of disease. PR is at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites.
Time Frame: From the first dose of study treatment to end of treatment response assessment (approximately 228 to 258 days)
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
percentage of participants | 82.0 [73.05 to 88.97]

3. Secondary Outcome: Complete Response (CR) Rate as Assessed by the Independent Review Facility (IRF) at the End of Treatment
Description: Complete response rate is defined as the percentage of participants with Complete Response (CR) according to the Revised Response Criteria for Malignant Lymphoma (Cheson et al., 2007). Disease response was evaluated by the IRF using CT scans, PET scans and pertinent clinical information. CR is the disappearance of all evidence of disease.
Time Frame: From the first dose of study treatment to end of treatment response assessment (approximately 228 to 258 days)
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
percentage of participants | 58.0 [47.71 to 67.80]

4. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the IRF at the End of Treatment
Description: Overall response rate was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) according to the Revised Response Criteria for Malignant Lymphoma (Cheson et al., 2007). Disease response was evaluated by the IRF using CT scans, PET scans and pertinent clinical information. CR is the disappearance of all evidence of disease. PR is at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites.
Time Frame: From the first dose of study treatment to end of treatment response assessment (approximately 228 to 258 days)
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
percentage of participants | 75.0 [65.34 to 83.12]

5. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator
Description: PFS was defined as the time from the date of the first dose of study treatment until the date of disease progression, relapse, or death from any cause.
Time Frame: From the first dose of study treatment to PFS assessment (up to 64 months)
Population: All participants. Patients who had not progressed, relapsed or died at the time of analysis were censored on the date of last valid disease assessment. If no tumor assessments were performed after the baseline visit, the patient was censored for PFS at the date after the first dose of study treatments.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
months | 48.3 [46.1 to 58.2]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as first occurrence of documented response (CR or PR) until the first occurrence of relapse or progression or death of any cause. CR: disappearance of all evidence of disease. PR: at least 50% regression of measurable disease compared to tumors measured by a baseline scan and no new sites.
Time Frame: From the response assessment to relapse, progression, or death (up to 64 months)
Population: All participants with data available. Participants who had not progressed, relapsed, or died at the time of analysis were censored for duration of response at the date of the last valid response assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 96
months | 45.6 [43.1 to 55.7]

7. Secondary Outcome: Percentage of Participants With Adverse Events as a Measure of Safety
Description: An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug or other protocol-imposed intervention. Preexisting conditions that worsened during the study were reported as adverse events.
Time Frame: From the first dose of study treatment to end of study (up to 5 years 4 months)
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
percentage of participants | 100.0

8. Secondary Outcome: Number of Participants With Grade 3 to 4 Infusion-Related (IRR) Adverse Events (AE) in Participants Receiving Shorter Duration Infusion (SDI)
Description: SDI 120 is a shorter duration infusion of 120 minutes and SDI 90 is shorter duration infusion of 90 minutes. Grade 3 IRR AE: Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae. Grade 4 IRR AE: Life-threatening consequences; urgent intervention indicated.
Time Frame: From the first dose of study treatment to end of treatment response assessment (approximately 228 to 258 days)
Population: Participants from the Safety population, all randomized participants who received at least 1 dose of study drug, who received shorter duration infusions.
Measure: Number; unit: participants
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 75
participants
  SDI 120 (n=5) | 0
  SDI 90 (n=70) | 0

9. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration Observed (Cmax) for Obinutuzumab
Description: Blood was collected for PK Parameters. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in micrograms per milliliter (μg/mL).
Time Frame: Cycle 1 Day 1 pre and post dose, Days 3,5, Day 8 pre and post-dose, Day 15 pre-dose. Cycle 8 Day 1 pre and post-dose, Days 5,8,12
Population: PK-Evaluable included all participants with viable PK data for analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
μg/mL
  Cycle 1 | 297 (110)
  Cycle 8 (n = 85) | 574 (183)

10. Secondary Outcome: Pharmacokinetics: Terminal Half-Life (t1/2) for Obinutuzumab
Description: T1/2 is the time required for the concentration of the drug to reach half of its original value. Blood was collected for PK Parameters. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in days
Time Frame: as for outcome 9
Population: PK-Evaluable included all participants with viable PK data for analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
days
  Cycle 1 (n = 37) | 6.04 (1.54)
  Cycle 8 (n = 21) | 23 (15.9)

11. Secondary Outcome: Pharmacokinetics: Clearance (Cl) for Obinutuzumab
Description: Cl is the volume of serum cleared of the drug per unit of time. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in milliliters/day (mL/day).
Time Frame: as for outcome 9
Population: PK-Evaluable included all participants with viable PK data for analysis.
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
mL/day
  Cycle 1 (n = 54) | 456 (254)
  Cycle 8 (n = 37) | 143 (59.8)

12. Secondary Outcome: Pharmacokinetics: Volume of Distribution (V) for Obinutuzumab
Description: V is the apparent volume in which a drug is distributed in the body. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in milliliters (mL).
Time Frame: as for outcome 9
Population: PK-Evaluable included all participants with viable PK data for analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
mL
  Cycle 1 (n = 54) | 4580 (2450)
  Cycle 8 (n = 37) | 9210 (17000)

13. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve 7 Day (AUC7day)
Description: Blood was collected for PK parameters. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA) measured in in day times micrograms per milliliter (day*μg/mL).
Time Frame: as for outcome 9
Population: PK-Evaluable included all participants with viable PK data for analysis.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Obinutuzumab + CHOP
Number analyzed (Participants) | 100
day*μg/mL
  Cycle 1 (n = 59) | 1320 (440)
  Cycle 8 (n = 74) | 3300 (1130)

14. Secondary Outcome: Pharmacodynamics: Peripheral Blood CD19-positive B-cell Count
Time Frame: Up to approximately 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment to clinical data cut-off: 23 December 2016 (up to 5 years, 4 months)
Description: All participants who received at least 1 dose of study drug.
Arm/Group | Obinutuzumab + CHOP
Serious Adverse Events (participants affected / at risk) | 38/100
Other Adverse Events (participants affected / at risk) | 100/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + CHOP (N=100)
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 2
Catheter site cellulitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Herpes zoster disseminated (Infections and infestations) | 1
Colonic abscess (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 14
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Acute left ventricular failure (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Spondylitic myelopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + CHOP (N=100)
Fatigue (General disorders) | 48
Chills (General disorders) | 41
Pyrexia (General disorders) | 26
Mucosal inflammation (General disorders) | 10
Oedema peripheral (General disorders) | 9
Chest pain (General disorders) | 7
Pain (General disorders) | 6
Asthenia (General disorders) | 5
Nausea (Gastrointestinal disorders) | 59
Diarrhoea (Gastrointestinal disorders) | 38
Vomiting (Gastrointestinal disorders) | 31
Constipation (Gastrointestinal disorders) | 29
Stomatitis (Gastrointestinal disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 5
Oral pain (Gastrointestinal disorders) | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 56
Skin abrasion (Injury, poisoning and procedural complications) | 5
Neuropathy peripheral (Nervous system disorders) | 24
Headache (Nervous system disorders) | 20
Dizziness (Nervous system disorders) | 17
Dysgeusia (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 40
Rash (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7
Night sweats (Skin and subcutaneous tissue disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 40
Anaemia (Blood and lymphatic system disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Urinary tract infection (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 6
Candida infection (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 5
Insomnia (Psychiatric disorders) | 14
Anxiety (Psychiatric disorders) | 10
Weight decreased (Investigations) | 12
Ejection fraction decreased (Investigations) | 5
Hypotension (Vascular disorders) | 15
Tachycardia (Cardiac disorders) | 9
Lacrimation increased (Eye disorders) | 5
Vision blurred (Eye disorders) | 5
Dysuria (Renal and urinary disorders) | 5
Haemorrhoids (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.